CLINICAL TRIAL: NCT04413149
Title: Observational Study of Clinical Features and Outcome of Interstitial Lung Disease With Anti-neutrophil Cytoplasmic Antibody in Chinese Patients.
Brief Title: Anti-neutrophil Cytoplasmic Antibody in Interstitial Lung Disease.
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-ANCA-positive ILD
Record Dates: First submitted 2020-05-25; First posted 2020-06-02 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Interstitial Lung Disease; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
Keywords: Interstitial Lung Disease; Anti-Neutrophil Cytoplasmic Antibody; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
MeSH Terms: conditions — Lung Diseases, Interstitial; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the clinical features and long-term outcome of anti-neutrophil cytoplasmic antibody (ANCA)-positive interstitial lung disease (ILD) and assess the difference between microscopic polyangiitis (MPA) associated ILD and isolated ANCA-positive idiopathic interstitial pneumonia.

DETAILED DESCRIPTION:
ILD patients with serum ANCA-positivity were enrolled in this study.

1. Baseline data collection:

   1. Demographics information (age, gender)
   2. Clinical course
   3. Clinical symptoms and signs (cough, dyspnea, fever, fatigue, crackling, clubbing fingers, mechanics hand)
   4. Laboratory findings (blood and urine routine, liver and renal function tests, erythrocyte sedimentation rate, C reactive protein)
   5. Serologic tests (ANA , Rheumatoid factor , Anti-cyclic citrullinated peptide (CCP), Anti-dsDNA, Anti-Ro (SS-A), Anti-La (SS-B), Anti-Smith, Anti-Scl-70, Anti-Jo-1)
   6. Systemic manifestation if diagnosed as systemic vasculitis
   7. Pulmonary function tests (ventilation and diffusion capacity test)
   8. Chest high-resolution computed tomography (HRCT)
2. Treatment: treatment will be given according to the experience of each pulmonologist.
3. Follow-up:

   1. Patients were followed up at least once a year and basic laboratory tests, serologic autoantibodies, pulmonary function test and chest HRCT were evaluated routinely
   2. Follow-up end point was April 2019.
4. Outcome

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged from 18 to 85 years with informed consent
* Have a diagnosis of ILD based on clinical symptoms and radiologic features, with or without histopathologic results
* Have available ANCA testing results during the first visit and follow-up period

Exclusion Criteria:

* Connective tissue disease associated ILD
* ILD induced by drug, environment, or occupational exposure
* Hypersensitivity pneumonitis and sarcoidosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interstitial lung disease patients with anti-neutrophil cytoplasmic antibody.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juhong Shi, M.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Sun X, Zhu W, Zhou C, Xue P, Li Z, Zhang W, Zhao J, Zhang T, Peng M, Shi J, Wang C. Clinical significance of anti-neutrophil cytoplasmic antibody in idiopathic interstitial pneumonia: a retrospective observational study. BMC Pulm Med. 2025 May 29;25(1):271. doi: 10.1186/s12890-025-03736-4. PMID 40442650

RESULTS

PARTICIPANT FLOW:
Groups:
- MPA-ILD Group: Among all the patients with ANCA-positive ILD, patients who fulfilled the MPA criteria were defined as MPA-ILD group.
- ANCA-IIP Group: Patients with isolated ANCA-positivity who did not fulfill the MPA criteria were classified as ANCA-IIP group.
Period: Overall Study
Arm/Group | MPA-ILD Group | ANCA-IIP Group
Started | 31 | 49
Completed | 20 | 44
Not Completed | 11 | 5
Not completed — Death | 10 | 5
Not completed — Lung transplantation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MPA-ILD Group | ANCA-IIP Group | Total
Number analyzed (Participants) | 31 | 49 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [47 to 67] | 59 [52 to 65] | 60 [51 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 12 | 24 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 31 | 49 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 31 | 49 | 80
Follow-up time [Median (Inter-Quartile Range); unit: months] | 36 [21 to 52] | 41 [28 to 64] | 40 [27 to 58]
Fever [Count of Participants; unit: Participants] | 16 | 10 | 26
Cough [Count of Participants; unit: Participants] | 28 | 42 | 70
Dyspnea [Count of Participants; unit: Participants] | 20 | 29 | 49
Fatigue [Count of Participants; unit: Participants] | 6 | 5 | 11
Arthralgia [Count of Participants; unit: Participants] | 8 | 15 | 23
Crackling sound [Count of Participants; unit: Participants] | 19 | 26 | 45
Rash [Count of Participants; unit: Participants] | 3 | 7 | 10
Clubbing fingers [Count of Participants; unit: Participants] | 5 | 2 | 7
Mechanics hand [Count of Participants; unit: Participants] | 0 | 2 | 2
Gottron's sign [Count of Participants; unit: Participants] | 1 | 2 | 3
Renal involvement [Count of Participants; unit: Participants] | 30 | 0 | 30
Nervous system involvement [Count of Participants; unit: Participants] | 3 | 0 | 3
Cardiovascular involvement [Count of Participants; unit: Participants] | 2 | 0 | 2
Retinal involvement [Count of Participants; unit: Participants] | 1 | 0 | 1
White blood cell [Median (Inter-Quartile Range); unit: ×10^9 cells/L] | 9.34 [7.15 to 13.56] | 7.44 [5.95 to 9.75] | 8.54 [6.18 to 10.36]
Neutrophil [Median (Inter-Quartile Range); unit: ×10^9 cells/L] | 6.79 [5.06 to 9] | 4.68 [3.76 to 6.94] | 5.65 [3.97 to 7.81]
Lymphocyte [Median (Inter-Quartile Range); unit: ×10^9 cells/L] | 1.47 [1.06 to 2.41] | 2 [1.55 to 2.33] | 1.90 [1.42 to 2.36]
Hemoglobin [Median (Inter-Quartile Range); unit: g/L] | 116 [95 to 139] | 137 [130 to 149] | 132 [116 to 147]
Platelet [Median (Inter-Quartile Range); unit: ×10^9 cells/L] | 251 [202 to 322] | 234 [176 to 284] | 246 [186 to 290]
Erythrocyte sedimentation rate [Median (Inter-Quartile Range); unit: mm/h] | 86 [49 to 99] | 28 [13 to 62] | 53 [17 to 87]
C reactive protein [Median (Inter-Quartile Range); unit: mg/dL] | 35.77 [5.67 to 71.18] | 13.87 [2.21 to 30.42] | 15.92 [3.88 to 53.70]
PaO2 [Median (Inter-Quartile Range); unit: mmHg] — PaO2: arterial oxygen tension
  mmHg | 71.5 [64.5 to 83] | 77.4 [72.3 to 82.2] | 75.9 [69.8 to 82.2]
Creatinine [Median (Inter-Quartile Range); unit: μmol/L] | 73 [61 to 104] | 67 [57 to 74] | 68 [57 to 79]
MPO-ANCA positive [Count of Participants; unit: Participants] — MPO: myeloperoxidase ANCA titres were measured by ELISA
  Participants | 26 | 19 | 45
PR3-ANCA positive [Count of Participants; unit: Participants] — PR3: proteinase 3 ANCA titres were measured by ELISA
  Participants | 0 | 2 | 2
Rheumatoid factor [Median (Inter-Quartile Range); unit: IU/mL] | 113.1 [53.5 to 207.8] | 26.7 [6.8 to 442.9] | 55.9 [22.7 to 211]
ANA positive [Count of Participants; unit: Participants] — ANA: antinuclear antibody
  Participants | 15 | 30 | 45
Anti-CCP positive [Count of Participants; unit: Participants] — Anti-CCP: anti-cyclic citrullinated peptide antibody
  Participants | 0 | 8 | 8
SSA positive [Count of Participants; unit: Participants] | 3 | 6 | 9
SSB positive [Count of Participants; unit: Participants] | 2 | 2 | 4
Jo-1 positive [Count of Participants; unit: Participants] — Jo-1: anti-Jo-1
  Participants | 0 | 1 | 1
Scl-70 positive [Count of Participants; unit: Participants] — Scl-70: anti-Scl-70
  Participants | 1 | 1 | 2
FEV1 [Mean (Standard Deviation); unit: percent predicted] — FEV1: forced expiratory volume in 1 s
  percent predicted | 79.36 (17.92) | 84.03 (16.93) | 82.35 (17.32)
FVC [Mean (Standard Deviation); unit: percent predicted] — FVC: forced vital capacity
  percent predicted | 78.30 (16.89) | 83.84 (19.10) | 81.85 (18.42)
TLC [Mean (Standard Deviation); unit: percent predicted] — TLC: total lung capacity
  percent predicted | 74.16 (12.73) | 79.53 (13.55) | 77.59 (13.43)
DLCO [Mean (Standard Deviation); unit: percent predicted] — DLCO: diffusing capacity of lung for carbon monoxide
  percent predicted | 56.56 (17.52) | 62.12 (14.09) | 60.12 (15.53)
Ground-glass opacity [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 25 | 44 | 69
Consolidation [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 4 | 4 | 8
Traction bronchiectasis [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 16 | 20 | 36
Honeycombing [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 11 | 8 | 19
Pulmonary artery dilation [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 3 | 1 | 4
Reticular pattern [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 20 | 29 | 49
Curved linear opacity [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 5 | 12 | 17
Pleural thickening [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 4 | 9 | 13
Interlobular septal thickening [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 16 | 23 | 39
Micronodular pattern [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 5 | 6 | 11
Subpleural bulla [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 10 | 10 | 20
Enlarged mediastinal lymph node [Count of Participants; unit: Participants] — performance in chest HRCT findings
  Participants | 2 | 3 | 5
Usual interstitial pneumonia [Count of Participants; unit: Participants] | 4 | 3 | 7
Nonspecific interstitial pneumonia [Count of Participants; unit: Participants] | 18 | 33 | 51
Unclassifiable HRCT pattern [Count of Participants; unit: Participants] | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Death From All Causes
Description: Death from all causes Retrieved from medical records.
Time Frame: From baseline until the date of death from all cause, up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | MPA-ILD Group | ANCA-IIP Group
Number analyzed (Participants) | 31 | 49
Participants | 10 | 5

2. Primary Outcome: Number of Patients Who Underwent Lung Transplantation
Description: Number of patients who underwent lung transplantation Retrieved from medical records.
Time Frame: From baseline until the date of transplantation, up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | MPA-ILD Group | ANCA-IIP Group
Number analyzed (Participants) | 31 | 49
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | MPA-ILD Group | ANCA-IIP Group
All-Cause Mortality (participants affected / at risk) | 10/31 | 5/49
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/49
Other Adverse Events (participants affected / at risk) | 0/31 | 0/49

LIMITATIONS AND CAVEATS:
Selection bias is possible due to its retrospective nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04413149/Prot_SAP_000.pdf